CLINICAL TRIAL: NCT01345487
Title: Effect of Protein From Animal and Vegetable Sources on Appetite
Acronym: PAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arne Astrup (Other)
Responsible Party: Sponsor-Investigator, Arne Astrup, M.D, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B275
Record Dates: First submitted 2011-04-27; First posted 2011-05-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Focus of Study: Appetite
Keywords: appetite; protein; legumes; meat
MeSH Terms: interventions — Plant Proteins, Dietary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Vegetable Protein (Other): Meal with 10 E% protein from fava beans/split peas
  Interventions: Other: Vegetable Protein
- High Vegetable protein (Experimental): Meal with 20 E% protein from fava beans/split peas
  Interventions: Other: Vegetable Protein
- High Animal Protein (Experimental): Meal with 20 E% protein from pork/beef
  Interventions: Other: Animal protein

INTERVENTIONS:
Other: Vegetable Protein — Vegetable protein in the form of fava beans/split peas
  Arms: High Vegetable protein; Low Vegetable Protein
Other: Animal protein — Protein in the form of minced pork/beef
  Arms: High Animal Protein

SUMMARY:
New Nordic diet guidelines advocate a reduction in consumption of protein from animal sources such as beef and pork, due to environmental concerns. Instead, intake of protein from vegetable sources such as legumes and pulses should be increased. However, little is known about the effect of protein from (Nordic grown) beans and peas on body weight and appetite regulation.

The objective of this study is to examine if protein from vegetable sources (beans and peas) is comparable to protein from animal sources regarding acute meal-induced satiety.

DETAILED DESCRIPTION:
Design:

Single-blind randomized 3-way crossover meal study

Subjects:

* 48 young healthy men (Age: 18-50 years; BMI: 19-30 kg/m2).
* Expected completers: n=42.

End points:

* Subjective appetite (VAS) (every 30 min for 3 hours)
* Ad libitum energy intake (3 hours after test meal)

Experimental diets:

Iso-caloric breakfast meals (3.5 MJ) with same energy density:

A. Fava beans + Split peas (20 protein E%) B. Fava beans + Split peas + potato (10 protein E%) C. Pork/beef + potato (20 protein E%)

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* 18-50 y
* body mass index (BMI) 18.5-30.0

Exclusion Criteria:

* smoking
* participation in other studies for 4 mo prior to entry
* weight gain/loss > 3 kg for to mo prior to entry
* Strenuous physical activity for > 10 h/wk
* Use of medication that can affect appetite
* food allergies or relevance for the test meals
* Psychiatric or metabolic disorders prohibiting participation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Composite appetite score area under the curve (180 min) | Assessed every 30 min for 180 min after each of the three test meals which are served 1 wk apart
  Composite score calculated from 10 cm visual analogue scale ratings:
  (desire to eat + hunger + prospective food consumption + (100-fullnes) + (100-satiety))/5
Ad libitum energy intake | Assessed 180 min after each of the 3 test meals, which are served 1 wk apart
  180 min after each test meal an ad libitum meal of spaghetti bolognese is served, and the total energy intake is recorded.

SECONDARY OUTCOMES:
Appetite ratings | Assessed every 30 min for 180 min after each or the 3 test meals which are served 1 wk apart
  Assessment of hunger, fulness, satiety, desire to eat and prospective food consumption from 10 cm visual analogue scale ratings every 30 min after meal consumption for 3 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Frederiksberg C, Denmark